CLINICAL TRIAL: NCT04355208
Title: Shade Evaluation of Monochromatic Versus Polychromatic Layering Techniques in Restoration of Fractured Incisal Angle: Randomized Controlled Trial
Brief Title: Shade Evaluation of Monochromatic Versus Polychromatic Layering Techniques Inrestoration of Fractured Incisal Angle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Badry Khalaf Hashem, Master degree studnet, Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3M™ Filtek™ Universal
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Anterior Teeth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Restoration of anterior teeth using monochromatic layering technique using body shade (filtek universal from 3m
  Interventions: Other: (3M™ Filtek™ Universal )
- comparator (Active Comparator): Restoration of anterior teeth using polychromatic layering technique using Enamel and Dentin shades (filtek Z350 xt from 3m
  Interventions: Other: (3M™ Filtek™ Universal )

INTERVENTIONS:
Other: (3M™ Filtek™ Universal ) — universal nanofillers resin composite (3M™ Filtek™ Universal )

SUMMARY:
This clincl trial will be conducted to compare theShade Evaluation of Monochromatic versus Polychromatic layering techniques in restoration of Fractured incisal angle

DETAILED DESCRIPTION:
The use of enamel and dentin shades allow us to reproduce anatomical features such as incisal edge translucency, halo effect, other internal colors and pigments such as craze lines, white patches, white horizontal striations .

Anterior composites usually have small filler particles to increase smoothness, nanotechnology has enabled recent advances in dental composite restorations. As a result , a different category of composite resins has emerged, known as nanocomposites.

However polychromatic layering is considered to be technique sensitive, from detection of details to proper reproduction of such fine details.

The presence of discrepancies between the classic shade guides and the actual shade of composite makes that task more difficult.

The use of monochromatic layering with only body shade can serve as a substitute for enamel and dentin, since it has an intermediate opacity between enamel and dentin , and can serve as an easier option with less technique sensitivity than polychromatic layering.

Filtek universal as claimed by the company manufacturer to have A "NaturalMatch" which is a term that describes the combination of 3M technologies and features present within 3M™ Filtek™ Universal restorative.

it contains nanofillers, pigments and proprietary low-stress monomers which gives Filtek™ Universal Restorative a combination of esthetic and universal opacity which in turn allow shade blending and making the restoration more invisible with surrounding dentition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with fractured incisal angle.
2. Vital teeth.
3. Anterior Permanent teeth.
4. Good oral hygiene.
5. Co-operative patients approving to participate in the study.

Exclusion Criteria:

1. Non vital teeth.
2. Severe or active periodontal disease.
3. Severe medical complications.
4. Uncooperative patients

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Shade matching | immediate after restoration
  shade matching using Modified USPHS Criteria and Visual inspection using Digital Photography